CLINICAL TRIAL: NCT01150019
Title: Correlation Between Circulating Resistin and Vascular Inflammation Measured by 18FDG-PET in Obese Person
Brief Title: Correlation Between Circulating Resistin and Vascular Inflammation Measured by 18F-fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) (18FDG-PET)
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Kyung Mook Choi, Korea University
Other Study IDs: PET_Resistin
Record Dates: First submitted 2010-06-09; First posted 2010-06-24 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-04

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; vascular inflammation; resistin; adiponectin; 18FDG-PET
MeSH Terms: conditions — Atherosclerosis | interventions — Cross-Sectional Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma, whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Obese Group
  Interventions: Other: Cross sectional study
- Non Obese Group
  Interventions: Other: Cross sectional study

INTERVENTIONS:
Other: Cross sectional study — This is not intervention study. The purpose of the study is to examine the relationship between various adipokine levels and PET imaging at the cross section setting

SUMMARY:
Vascular inflammation is a key factor in both the pathogenesis and outcome of atherosclerosis.Resistin was shown to induce vascular endothelial dysfunction and vascular smooth muscle cell proliferation.

18F-fluorodeoxyglucose (FDG) positron emission tomography (PET) is a promising tool for identifying and quantifying vascular inflammation within atherosclerotic plaques.Therefore, the purpose of the study is to demonstrate the correlation between circulating resistin and vascular inflammation detected by 18FDG-PET in obese persons.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers for visiting routine medical check in our clinic

Exclusion Criteria:

* History of cardiovascular disease (myocardial infarction, unstable angina,stroke, or cardiovascular revascularization)
* Diabetes
* Hypertension
* Malignancy
* Severe renal or hepatic disease
* Subjects taking medications that might affect inflammation such as non-steroidal anti-inflammatory drugs (NSAIDs) and statin

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participats who underwent a medical health check in the health promotion center in Korea Guro University
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Vascular inflammation in carotid arterial wall represented as the target-to-background ratio (TBR) using FDG-PET | 12 weeks

SECONDARY OUTCOMES:
Circulating serum adiponectin levels | 12 weeks
carotid intima-media thickness levels measured using ultrasonography | 12 weeks
Circulating serum resistin levels | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mook Choi, MD.PhD, Principal Investigator — Korea University
Locations (1):
- Hae Yoon Choi, Seoul, South Korea